CLINICAL TRIAL: NCT07071454
Title: Preventing Early-Onset Colorectal Cancer in the VA Using a Multilevel Screening Intervention
Brief Title: Preventing Early-Onset Colorectal Cancer in the VA
Acronym: PRECISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: IIR 23-005
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Neoplasms; Mass Screening
Keywords: early onset colorectal cancer; risk stratification; behavioral intervention
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The investigators will use a electronic health record (EHR) based risk score, which has been previously validated, to prospectively identify high-risk and non-high-risk individuals for a multilevel (patient, provider, and clinic) screening intervention. The investigators will employ a 2x2 factorial design for the patient and provider level interventions to quantify independent and potentially synergistic effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Patient intervention (Experimental): Only patients receive intervention
  Interventions: Behavioral: Patient intervention
- PCP intervention (Experimental): Only PCP receives intervention
  Interventions: Behavioral: PCP intervention
- Combined (Experimental): Both patient and PCP receive intervention
  Interventions: Behavioral: Patient intervention; Behavioral: PCP intervention
- Control (No Intervention): Neither patient nor PCP receives intervention

INTERVENTIONS:
Behavioral: Patient intervention — Patient intervention has 2 components. 1) The investigators will send patients a letter that promotes screening and contains targeted messages based on the individual's demographic characteristics. 2) Study staff who is trained in patient navigation will call each patient up to 3 times to confirm receipt of the letter and conduct one-on-one education about screening using a standardized script.
  Arms: Combined; Patient intervention
Behavioral: PCP intervention — PCP intervention has 2 components. 1) PCPs of patients who are randomized to this group will receive an initial email that provides a list of all patients assigned to the PCP who are randomized to the PCP intervention. PCPs will be specifically informed which patients are high-risk. The email will also include a personal report card with the percentage of patients assigned to the provider who are up-to-date with CRC screening in two age groups: 45-49 years and 50-75 years. Subsequently, PCPs will receive weekly emails with a list of patients randomized to the PCP intervention who are scheduled for a clinic visit with them. 2) The investigators will design a local clinical dashboard using Microsoft Power BI that allows PCPs to view a list of their patients who are randomized to the PCP intervention as well as provide a link to this in each email. High-risk patients will be specifically marked.
  Arms: Combined; PCP intervention

SUMMARY:
Colorectal cancer is a leading cause of cancer death among Veterans. The starting age for colorectal cancer screening has been lowered from 50 to 45 years in response to the rising incidence of early-onset colorectal cancer (EOCRC), but how to best engage younger Veterans in screening is unclear. The investigators will 1) develop and validate a novel risk score for EOCRC derived from the VA electronic health record data, 2) conduct a multilevel screening intervention that targets individuals aged 45-49 years and informs high-risk individuals and their providers about their risk status for EOCRC, and 3) determine barriers and facilitators to implementing the intervention using a qualitative process evaluation. Aim 2 is the focus of the trial. The overall goal of this study is to create and test a risk stratification approach to prevent EOCRC, which may be especially useful for younger individuals who are less likely to participate in preventive care.

DETAILED DESCRIPTION:
Background: Incidence and mortality of early-onset colorectal cancer (EOCRC), defined as colorectal cancer (CRC) diagnosed before age 50 years, has been increasing in the US since the 1990s. In response to these concerning trends, in 2021 the US Preventive Services Task Force recommended lowering the age to initiate CRC screening from 50 to 45 years. Within the VA health care system, 60% of eligible individuals aged 50-75 years and only 42% of those aged 45-49 years were up-to-date with screening in May 2024. Younger individuals are less likely to perceive the need for screening, but informing individuals who are at higher risk about their status may increase their interest and participation in screening.

Significance: CRC is a leading cause of cancer death among Veterans. To maximize CRC screening benefit in individuals younger than 50 years, it is critical to 1) identify high-risk individuals in this age group who may be targeted for screening and 2) assess the effectiveness and implementation of interventions to promote screening in all younger individuals. Innovation & Impact: Currently there are no risk scores for EOCRC in clinical use, and risk scores developed for research often use genetic and survey data but omit more readily accessible information from the electronic health record (EHR) to identify individuals at increased risk. In addition to identifying high-risk individuals, it is also crucial to study interventions that will increase screening in the younger population. Otherwise, data show that younger adults are less likely to engage in screening and passive adoption of new clinical guidelines occurs slowly among physicians.

Specific Aims:

Aim 1: To develop and validate a risk score for EOCRC using EHR data Aim 2: To determine the effectiveness of a multilevel intervention to increase screening in individuals aged 45-49 years, using personal risk as a motivator for high-risk individuals. This aim is the focus of the trial.

Aim 3: To evaluate the implementation of the multilevel intervention.

Methodology: The investigators plan to 1) build and validate an EOCRC risk score using EHR data from the VA Corporate Data Warehouse (CDW), 2) identify a prospective cohort of Veterans aged 45-49 years and conduct a 2x2 factorial multilevel intervention that includes informing high-risk patients and their primary care providers about their risk status, and 3) assess for barriers and facilitators to implementing the multilevel intervention through a qualitative process evaluation with key informants.

Next Steps/Implementation: If this novel risk stratification strategy to prevent EOCRC is effective at a single site, then the investigators will work with partners to implement it throughout the VA and test it outside of the VA system.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-49 years at screening

Exclusion Criteria:

* Up-to-date with CRC screening based on the USPSTF guideline (e.g., colonoscopy within the past 10 years or FIT within the past year)
* Prior CRC diagnosis
* Prior total colectomy
* Limited life expectancy (defined as terminal illness, hospice enrollment, or documented life expectancy <6 months on the medical problem list or a health factor in the EHR
* Deactivated national CRC screening and surveillance reminder (due to risk level or comorbidities)

Ages: 45 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 536 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Screening participation rate in groups that received vs. did not receive the patient intervention | 6 months
  For the patient intervention analysis, the investigators will compare the patient and combined arms vs. the PCP and control arms. Completion of FIT, colonoscopy, and any other USPSTF-recommended screening test will be considered to meet the outcome.
Screening participation rate in groups that received vs. did not receive the PCP intervention | 6 months
  For the PCP intervention analysis, the investigators will compare the PCP and combined arms vs. the patient and control arms. Completion of FIT, colonoscopy, and any other USPSTF-recommended screening test will be considered to meet the outcome.

SECONDARY OUTCOMES:
Screening participation rate in high-risk vs. non-high-risk individuals | 6 months
  Of the 536 individuals the investigators plan to enroll in the trial, 536*(3/4)=402 will be randomized to one of the three intervention arms. The investigators will compare high- vs. non-high-risk individuals in the intervention arms (n=201 in each arm).

OTHER OUTCOMES:
Screening participation rate in individual groups | 6 months
  The investigators will compare screening uptake a) in the combined patient/PCP intervention arm vs. the single-intervention arm with higher uptake and b) in the single-intervention arm with lower uptake vs. the control arm
Screening participation rate in Black vs. non-Black individuals | 6 months
  The investigators will compare screening uptake in the three intervention arms for Black vs. non-Black individuals.
Shared decision making in different intervention groups | 6 months
  The investigators will compare shared decision-making (SDM)-measured by the SDM Process scale-in arms that received a) the patient intervention and b) the PCP intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Liang, MD MPH, Principal Investigator — VA NY Harbor Healthcare System, New York, NY
Locations (1):
- VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No